CLINICAL TRIAL: NCT06031246
Title: Selective Lymph Node Dissection for cT1N0M0 Invasive Non-small Cell Lung Cancer With CTR>0.5 Located in the Apical Segment: a Single-arm, Multi-center, Phase III Trial
Brief Title: Selective Lymph Node Dissection for cT1N0M0 Invasive NSCLC With CTR>0.5 Located in the Apical Segment (ECTOP-1018)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Director in the Department of Thoracic Surgery, FUSCC, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SELLAS
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Lung Adenocarcinoma; Lymph Node Metastasis
MeSH Terms: conditions — Adenocarcinoma of Lung; Lymphatic Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Selective Lymph Node Dissection (Experimental): Selective Lymph Node Dissection is performed for cT1N0M0 Invasive Non-small Cell Lung Cancer With CTR>0.5 Located in the Apical Segment
  Interventions: Procedure: Selective Lymph Node Dissection

INTERVENTIONS:
Procedure: Selective Lymph Node Dissection — For patients with NSCLC with CTR>0.5 located in the apical segment, the inferior mediastinal lymph node was not need to dissected

SUMMARY:
This is a clinical trial from Eastern Cooperative Thoracic Oncology Project (ECTOP), numbered as ECTOP-1018. The goal of this clinical trial is to confirm the theraputic effect of selective lymph node dissection for cT1N0M0 invasive non-small cell lung cancer with CTR>0.5 located in the apical segment. The main questions it aims to answer are:

The 5-year overall survival of patients having cT1N0M0 invasive non-small cell lung cancer with CTR>0.5 located in the apical segment; The post-operative lymph node metastasis and recurrence-free survival. Participants will receive selective lymph node dissection as the surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who sign the informed consent form and are willing to complete the study according to the plan;
2. Aged from 18 to 80 years old;
3. ECOG equals 0 or 1;
4. Not receiving lung cancer surgery before;
5. Resectable peripheral cT1N0M0 tumors with CTR>0.5 located in the apical segment;
6. Non-lepidic predominant invasive NSCLC dignosed by frozen section;
7. Not receiving chemotherapy or radiotherapy before.

Exclusion Criteria:

1. Not cT1N0M0;
2. Nodules not located in the apical segment or CTR≤0.5;
3. Pre-invasive lung adenocarcinoma, lepidic predominant adenocarcinoma, or not lung adenocarcinoma diagnosed cytologically or pathologically;
4. Receiving lung cancer surgery before;
5. Receiving radiotherapy or chemotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 634 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
5-year overall survival | 5 years
  The event is defined as the death due to any causes.

SECONDARY OUTCOMES:
Lymph node metastasis | 5 years
  the lymph node metastasis situation of each pathological subtype
5-year recurrence-free survival | 5 years
  The event is defined as the tumor recurrence.
The accuracy of frozen section | 5 years
  The concordance of frozen section and final pathological diagnosis for invasiveness

CONTACTS AND LOCATIONS:
Overall Officials: Haiquan Chen, M.D., Principal Investigator — Fudan University
Locations (1):
- Chaoqiang Deng, Shanghai, Please Select, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Y, Deng C, Luo X, Yu Y, Zhang Y, Chen H. Protocol of a single-arm, multicenter, phase III trial for selective lymph node dissection in cT1N0M0 invasive non-small cell lung cancer with consolidation-tumor ratio >0.5 located in the apical segment: Eastern Cooperative Thoracic Oncology Projects ECTOP-1018 (SELLAS study). J Thorac Dis. 2024 Nov 30;16(11):8142-8148. doi: 10.21037/jtd-24-1114. Epub 2024 Nov 21. PMID 39678839